CLINICAL TRIAL: NCT01726998
Title: Effects of Locomotion Training With Assistance of a Robot-Driven Gait Orthosis in Hemiparetic Patients After Subacute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2012-0005
Record Dates: First submitted 2012-11-07; First posted 2012-11-15 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Stroke; Hemiparetic Patients After Subacute Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lokomat Group (Experimental)
  Interventions: Other: Robot-assisted gait therapy
- conventional gait training group (Active Comparator)
  Interventions: Other: conventional gait training

INTERVENTIONS:
Other: Robot-assisted gait therapy — Two groups received 30 minutes conventional gait training including Neurodevelopmental Treatment(NDT) basically. Robot-assisted gait therapy for 30 minutes with Lokomat® (Hocoma, Zurich, Switzerland) daily for 4 weeks, and the conventional gait training group received additional daily conventional gait training with NDT for the same periods.
  Arms: Lokomat Group
Other: conventional gait training — Two groups received 30 minutes conventional gait training including Neurodevelopmental Treatment(NDT) basically. Robot-assisted gait therapy for 30 minutes with Lokomat® (Hocoma, Zurich, Switzerland) daily for 4 weeks, and the conventional gait training group received additional daily conventional gait training with NDT for the same periods.
  Arms: conventional gait training group

SUMMARY:
The investigators aimed in this study to investigate the effects of 4 weeks robot-assisted locomotor training on motor recovery of lower extremities and walking ability compared with the conventional gait training in subacute post-stroke non-ambulatory hemiplegic patients.

72 first-ever stroke patients who could not walk independently (FAC < 2), and suffered within 6 months were enrolled and randomly assigned into 2 groups. The subjects with congestive heart failure, malignancies, cardiopulmonary dysfunctions, and who could not walk independently before stroke attack were excluded.

Two groups received 30 minutes conventional gait training including Neurodevelopmental Treatment (NDT) basically. The robotic assisted locomotor training group received additional robotic-assisted gait therapy for 30minutes with Lokomat® (Hocoma, Zurich, Switzerland) daily for 4 weeks, and the conventional gait training group received additional daily conventional gait training with NDT for the same periods. The independent walking ability(FAC ≥ 3), Functional Ambulation Category (FAC), Motricity index (MI), Fugl-Meyer assessment (FMA), Modified Barthel Index (MBI), Medical Research Council (MRC) for each lower extremity muscles were assessed before, during (2weeks) and after training. And the independent walking ability were followed until 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Hemiparesis as result of 1st stroke
2. No other neurologic or orthopedic disorder
3. Independent ambulation before the stroke
4. No severe medical illnesses
5. Hemiparesis: lower extremity strength graded ≤ 3 in more than 2 muscle groups
6. Functional ambulation classification (FAC) ≤ 1 : indicating a need for personal assistance in ambulation
7. The interval between stroke and start of the treatment
8. Time since stroke onset < 6 months
9. age: 20-80yrs old

Exclusion Criteria:

1. Unstable fractures
2. Severe osteoporosis
3. Severe skin problems
4. Severe joint problems
5. Major difference in leg length,
6. Body weight over 130 kg,
7. Orthostatic circulatory problem
8. Severe cognitive impairment

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
change of functional ambulation category point | baseline, during training (2weeks), post training (4weeks) & followed for 2months after training
  FAC is a functional walking test that evaluates ambulation ability. This is an 6-point scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, Seoul, South Korea